CLINICAL TRIAL: NCT02021981
Title: Improving Health Outcomes: Blood Pressure Program in Practice Sites Located in the Chicago Metropolitan Area and in Maryland
Brief Title: Improving Health Outcomes: Blood Pressure
Acronym: IHO:BP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: American Medical Association (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Omar Hasan, MBBS, MPH, MS, FACP, Vice President, Improving Health Outcomes, American Medical Association
Other Study IDs: #2013-1094
Record Dates: First submitted 2013-12-17; First posted 2013-12-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension
Keywords: Quality Improvement; Primary Care; Blood Pressure, High; Feedback; Knowledge
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Observational Group 1: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 2: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 3: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 4: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 5: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 6: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 7: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 8: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 9: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.
- Observation Group 10: Coach care teams in the practice site on how to implement evidence-based enhancements in hypertension care delivery processes, using established quality improvement principles and methods. In one year, figure out the best way to help different types of ambulatory clinical practices achieve improved blood pressure control.

SUMMARY:
This quality improvement project is focused on improving hypertension care delivery processes in ambulatory clinical practices, 5 in Illinois and 5 in Maryland for a total of 10 practice sites.The primary aim of this quality improvement project is to improve blood pressure control among patients receiving routine care for hypertension in a diverse group of ambulatory clinical practices. A secondary aim is for American Medical Association (AMA) and Johns Hopkins Medicine (JHM) quality improvement staff to figure out the best way to help clinical practices in achieving improved blood pressure control, including working to increase the use of home blood pressure monitoring.

ELIGIBILITY:
The Practice Sites must

* Self-identify as either primary care internal medicine, family practice, or cardiology
* Have an electronic health record
* Serve patient populations that are diverse and representative of the U.S. adult population
* Have a significant number of male and female patients, age 18 or older, voluntarily receiving care for hypertension
* Have the resources, staff, and commitment to complete this quality improvement project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This quality improvement project will be conducted in 10 ambulatory practice sites that are distinguished by their medical specialty and practice size. There are 9 diverse sites that specialize in family medicine and internal medicine. One site is a cardiology practice. Practices range in size from a mid-size medical group to a single-physician practice. The total number of physicians participating in this project is between 40 and 50. The sites are located in various neighborhoods in the Chicago and Baltimore metropolitan areas and in rural Maryland. The patient populations of the sites are representative of the United States population.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Improve blood pressure control | One year
  The primary aim of this quality improvement project is to improve blood pressure control among patients receiving routine care for hypertension in a diverse group of ambulatory clinical practices. Specifically, we will measure change from baseline in Systolic Blood Pressure at 12 months.

SECONDARY OUTCOMES:
The best way to help clinical practices improve blood pressure control | One year
  A secondary aim is for AMA and JHM quality improvement staff to figure out the best way to help clinical practices in achieving improved blood pressure control. Specifically, we will measure success in implementing changes in hypertension care delivery processes by surveying clinical practice staff.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Hasan, MBBS MPH FACP, Principal Investigator — American Medical Association
Locations (1):
- American Medical Association, Chicago, Illinois, United States